CLINICAL TRIAL: NCT02019355
Title: The Role of Calcipotriol in Treatment of Pre-cancerous Skin Lesions
Brief Title: Actinic Keratosis Study
Acronym: AK
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Lynn Cornelius, MD, Chief, Division of Dermatology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201303070
Record Dates: First submitted 2013-12-10; First posted 2013-12-24 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2013-12

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Fluorouracil; calcipotriene; Ointments; Petrolatum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- calcipotriol plus 5-fluorouracil (Experimental): calcipotriol 0.005% ointment and 5-fluorouracil 5% cream are mixed at 1:1 weight ratio. The compounded medication is applied topically twice a day for 4 days.
  Interventions: Drug: 5-fluorouracil 5% cream; Drug: Calcipotriol 0.005% ointment
- 5-fluorouracil plus vaseline (Active Comparator): 5-fluorouracil 5% cream and vaseline are mixed at 1:1 weight ratio. The compounded medication is applied topically twice a day for 4 days.
  Interventions: Drug: 5-fluorouracil 5% cream; Drug: Vaseline

INTERVENTIONS:
Drug: 5-fluorouracil 5% cream
  Other Names: Efudex
Drug: Calcipotriol 0.005% ointment
  Other Names: Calcipotriene; Dovonex; MC 903
  Arms: calcipotriol plus 5-fluorouracil
Drug: Vaseline
  Arms: 5-fluorouracil plus vaseline

SUMMARY:
The main purpose of this study is to determine the effectiveness of a new combination therapy for actinic keratosis. This study investigates a new indication for an FDA-approved topical medication, calcipotriol, for treatment of actinic keratosis, including how well it works and how safe it is when used in combination with the standard of care medication (5-fluorouracil) for the skin condition.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 50 years
* Presence of four to fifteen clinically typical, visible, and discrete actinic keratoses in 25 cm2 on any of the four anatomical sites: scalp, face, right upper extremity and left upper extremity
* Ability and willingness of the patient to participate in the study (Informed consent is obtained)

Exclusion Criteria:

* Treatment area is within 5 cm of an incompletely healed wound or a suspected basal-cell or squamous-cell carcinoma
* Treatment area contained hypertrophic and hyperkeratotic lesions, cutaneous horns, or lesions that had not responded to repeated cryotherapy
* Recent (within a month) use of medications that could interfere with evaluation of the treatment area (e.g., topical medications, artificial tanners, immunosuppressive medications, immunomodulating agents, cytotoxic drugs, ultraviolet B phototherapy, other therapies for actinic keratoses, or oral retinoids)
* Premenopausal Women (to avoid any risk of pregnancy)
* History of hypercalcemia or clinical evidence of vitamin D toxicity

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2013-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
percentage of change in the number of actinic keratoses from baseline | 8 weeks
  To compare the efficacy of topical 5-fluorouracil+calcipotriol vs. 5-fluorouracil alone in treatment of actinic keratosis in patients with multiple actinic keratoses at each of the four anatomical sites (scalp, face, right upper extremity and left upper extremity). The outcome of interest is percentage change from baseline number of actinic keratoses in the target treatment area on scalp, face, right upper extremity and left upper extremity at 8 weeks after treatment.

SECONDARY OUTCOMES:
complete and partial (>75%) clearance of actinic keratoses | 8wks
  o To determine complete and partial (>75%) clearance of actinic keratoses at 8 weeks after treatment.
Composite score of erythema, itching and skin pain after topical 5-fluorouracil+calcipotriol vs. 5-fluorouracil alone treatment of actinic keratoses | 4days
  To determine the composite scores of erythema, itching and pain (determined using standardized scales) following topical application of 5-fluorouracil+calcipotriol vs. 5-fluorouracil alone at the end of the 4-day treatment period.
Induction of TSLP expression in keratinocytes by calcipotriol | 4 days
  To examine the induction of TSLP expression in keratinocytes by calcipotriol at the site of the actinic keratoses at the end of 4-day treatment of course.
differences in response to topical 5-fluorouracil+calcipotriol vs. 5-fluorouracil alone between the four anatomical sites | 8wks
  To determine any differences in response to topical 5-fluorouracil+calcipotriol vs. 5-fluorouracil alone between the four anatomical sites at 8 weeks after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Cornelius, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Cunningham TJ, Tabacchi M, Eliane JP, Tuchayi SM, Manivasagam S, Mirzaalian H, Turkoz A, Kopan R, Schaffer A, Saavedra AP, Wallendorf M, Cornelius LA, Demehri S. Randomized trial of calcipotriol combined with 5-fluorouracil for skin cancer precursor immunotherapy. J Clin Invest. 2017 Jan 3;127(1):106-116. doi: 10.1172/JCI89820. Epub 2016 Nov 21. PMID 27869649